CLINICAL TRIAL: NCT06178874
Title: Insulin Degludec vs Insulin Glargine for Glycemic Control in Critical Illness Hyperglycemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Adham Haggag, Associate proffesor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R322/2023
Record Dates: First submitted 2023-11-18; First posted 2023-12-21 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Glycemic Control; Insulin; Critical Illness
MeSH Terms: conditions — Insulin Resistance; Critical Illness | interventions — Insulin Glargine; insulin degludec; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group S (Active Comparator): The random blood sugar in the patients in group S will be managed using regular insulin based on a sliding scale together with an Insulin Glargine, 0.2 units/kg , SC, initially to be titrated as per the clinical situation to be given at 9 PM
  Interventions: Drug: Insulin Glargine; Drug: Insulin regular
- Group L (Active Comparator): The random blood sugar in the patients in group L will be managed using regular insulin based on a sliding scale together with an Insulin Degludec 0.2 units/kg, SC, initially to be titrated as per the clinical situation to be given at 9 PM
  Interventions: Drug: Insulin Degludec; Drug: Insulin regular
- Group R (Active Comparator): The random blood sugar in the patients in group R will be managed using regular insulin based on a sliding scale
  Interventions: Drug: Insulin regular

INTERVENTIONS:
Drug: Insulin Glargine — hyperglycemic control
  Arms: group S
Drug: Insulin Degludec — hyperglycemic control
  Arms: Group L
Drug: Insulin regular — hyperglycemic control

SUMMARY:
The role of ultralong insulin in the control of the blood glucose level in diabetic patients is well known, the current study will discuss the role of ultralong insulin in controlling of hyperglycaemia in critical illness defined as failure or impending failure of an organ

DETAILED DESCRIPTION:
A standard monitor will be attached to the patients including 5 leads ECG, pulse oximeter, NIBP and IV line will be secured. The hemodynamic parameters will be recorded every 15 minutes.

The random blood sugar in the patients in group S will be managed using regular insulin based on a sliding scale as in Table 1 together with an Insulin Glargine, 0.2 units/kg , SC, initially to be titrated as per the clinical situation to be given at 9 PM.

The random blood sugar in the patients in group L will be managed using regular insulin based on a sliding scale as in table 1 together with an Insulin Degludec 0.2 units/kg, SC, initially to be titrated as per the clinical situation to be given at 9 PM.

The random blood sugar in the patients in group R will be managed using regular insulin based on a sliding scale THE total dose of insulin will be monitored, episodes of hypoglycaemia ' decrease of blood sugar less than 60gm/dl, the length of the hospital stay, the serum potassium level , the incidence of infection as evidenced by increase WBC or clinical evidence of infection, incidence of diabetic ketoacidosis and the incidence of acute kidney risk as evidenced by decrease of urine output < 0.5 ml/kg/hr for more than 6 hr and/or increase of the serum creatinine 1.5-2 times the baseline of Acute kidney injuries as evidenced by decrease of urine output < 0.5 ml/kg/hr for more than 12 hr and/or increase of the serum creatinine 2-3 times the baseline.

The CBC, Kidney function test, liver enzymes, serum creatinine, s.Na+, s.K+ , s.albumin, RBS will be collected on admission and every three days if there is no indication for close monitoring. Glycated haemoglobin will be collected once.

The blood sugar will be checked hourly using finger prick test and the glucose variabilities will be monitored.

Action for Hypoglycaemia: [18]

Mild (Adults who are conscious, orientated and able to swallow):

Check ABCDE, stop IV insulin Give 15-20g of quick acting carbohydrate, such as 5-7 sugar canned tablets or 150-200ml pure fruit juice. Test blood glucose level after 10-15 minutes and if still less than 70 mg/dl repeat treatment as above up to 3 times. If still hypoglycaemic, IV dextrose will be given

Moderate (Person conscious and able to swallow, but confused, disorientated or aggressive):

Check ABCDE, stop IV insulin. If capable and cooperative, treat as for mild hypoglycaemia. If not capable and cooperative but can swallow give 2 tubes of 40% glucose gel (squeezed into mouth between teeth and gums). Test blood glucose level after 10-15 minutes and if still less than 70mg/dl repeat as above up to 3 times. If still hypoglycaemic, consider IV dextrose or IM glucagon as per "severe" pathway Severe (Person unconscious/fitting or very aggressive or nil by mouth (NBM)) Check ABCDE, stop IV insulin. Give 100ml 20% dextrose or 200ml 10% dextrose over 15 minutes. Recheck glucose after 10 minutes and if still less than 70mg/dl, repeat treatment as above.

For all degrees of hypoglycaemia:

* once glucose > 70 mg/dl, and the patient is able to swallow, 20 gm of long-acting carbohydrates (two biscuits, slice of bread, 200-300ml milk) will be given, and if the patient is not able to swallow or NBM, 10% glucose infusion at 100ml/hr will be given until no longer NBM.
* once glucose > 70 mg/dl, intravenous regular insulin will be resumed at a rate 0.5U/hour for all groups and for group L and S, there will be reduction 20-30% in the next subcutaneous long-acting insulin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Blood glucose level >250 mg/dl for more than 24 h

Exclusion Criteria:

* Age less than 18 or greater than 60 years
* Diabetic Ketoacidosis
* Patients with recurrent episodes of hypoglycaemia-* Stress hyperglycemia
* Patients refusing to participate in the study.
* Patients with renal insufficiency
* Patients on corticosteroids

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-25 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
hyperglycemic control | 10 days of ICU stay
  the insulin dose needed for achievement of the glycemic goals by insulin degludec vs insulin Glargine in critically ill patient.

SECONDARY OUTCOMES:
length of ICU stay | from admission till discharge from ICU through a period of 2 weeks
  the effect of using long acting insulin on the length of icu stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt